CLINICAL TRIAL: NCT06708351
Title: Enhancing Cervical Cancer Screening and Treatment in Women Living With HIV in Kenya (ENHANCE LINKAGE)
Brief Title: Enhancing Cervical Cancer Screening and Treatment in Women Living With HIV in Kenya, the ENHANCE LINKAge Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael H Chung, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00008289; U01CA275120-01A1 (NIH); NCI-2024-08623 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EU6378-24 (Other: Emory University Hospital/Winship Cancer Institute); STUDY00008289 (Other: Emory University/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: HIV Infection; Human Papillomavirus-Related Cervical Carcinoma; Screening Strategy
MeSH Terms: conditions — HIV Infections | interventions — Practice Guidelines as Topic; Standard of Care; Health Promotion; Educational Status

STUDY DESIGN:
Intervention Model Description: hybrid type 2 implementation-effectiveness cluster randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aim 2, Arm I (ENHANCE LINKAge) (Experimental): Patients receive HPV self-testing kit and instruction on how to perform HPV self-testing on study. Patients undergo vaginal self-swab and receive results by text message. Patients also receive mobile text message reminders for triage or treatment for women that test positive with HPV.
  Interventions: Other: Health Promotion and Education; Procedure: HPV Self-Collection; Other: Text Message-Based Navigation Intervention
- Aim 2 (standard care) (Active Comparator): Patients undergo standard of care at clinics that have VIA testing
  Interventions: Other: Best Practice

INTERVENTIONS:
Other: Best Practice — Receive standard care
  Other Names: standard of care; standard therapy
  Arms: Aim 2 (standard care)
Other: Health Promotion and Education — Receive instructions on how to use HPV self-testing kit
  Arms: Aim 2, Arm I (ENHANCE LINKAge)
Procedure: HPV Self-Collection — Undergo HPV self-collection
  Other Names: At-home HPV Self Collection; HPV Self Collection; Human Papillomavirus Self-Collection
  Arms: Aim 2, Arm I (ENHANCE LINKAge)
Other: Text Message-Based Navigation Intervention — Receive text messages for HPV testing results and triage and treatment reminders
  Other Names: Automated Text Message-Based Navigation; Text Message-Based Navigation
  Arms: Aim 2, Arm I (ENHANCE LINKAge)

SUMMARY:
Background In sub-Saharan Africa (SSA), human papillomavirus (HPV) and HIV create a dual burden of disease that causes significant morbidity and mortality in the form of cervical cancer (CC). Women living with HIV (WLWH) have a six-fold higher risk of developing precancerous lesions that persist and progress to CC, which is the leading cause of cancer mortality among women in Kenya. Significant support from the Go Further campaign, represented by donors such as the President's Emergency Plan for AIDS Relief (PEPFAR), the George W. Bush Institute, UNAIDS, Merck, and Roche, to integrate CC screening into HIV clinics represents an exceptional opportunity to scale CC impact across SSA, but only if implementation science evidence is available to inform strategy. Currently, the impact of Go Further has been undermined by fractured linkages to care and insensitive screening methods; in Kenya, less than 2% of WLWH screened have received appropriate treatment. Implementation science studies are needed to better understand and surmount barriers to integrated care in publicly funded HIV clinics.

Broad objective This study seeks to explore and innovate strategies to overcome patient-, provider-, and system-level barriers to implementing CC screening and referral guidelines, link WLWH who require further diagnostic testing and/or treatment with effective and accessible care, and document services for accountability and quality improvement. In this proposal, our team will apply our extensive implementation science expertise and partnerships with Kenya Ministry of Health (MOH) to adapt and test evidence-based strategies (e.g., HPV self-testing, care navigators, and the WEMA mHealth app [tested and scaled in Tanzania]) that address key multi-level barriers identified through a formative, stakeholder-engaged research phase.

Methodology Using the EPIS framework to guide our project, we will: Aim 1a), Explore (engage a multi-disciplinary stakeholder advisory board to co-design the intervention package and prioritize implementation strategies that align with local capacity, opportunities, and motivations; Aim 1b), Prepare (develop tools and strengthen capacity at clinics to implement the strategies; Aim 2), Implement and evaluate the package of implementation strategies via a cluster-randomized stepped wedge trial in 9 clinics (assessing implementation [provision of CC screening with HPV self-testing] and effectiveness [proportion of HPVpositive WLWH who receive subsequent diagnostic triage and/or treatment] over months 0-12; and Aim 3), assess Sustainability (costs, cost-effectiveness, and transfer of delivery from study to local staff over months 13-18.

Significance of the study The overall goal of this study is to employ rigorous empirical methods to adapt and test implementation strategies that expand the scope of HIV care to screen for and treat early precancerous CC lesions in a sustainable, scalable way. Through partnering with Kenya's MOH, this project will have critical institutional support and dissemination capability, and will directly inform public health practice and policy.

DETAILED DESCRIPTION:
Broad Objectives This study seeks to inform the effective and sustainable integration of early detection and successful treatment of precancerous cervical lesions among women living with HIV (WLWH) ages 25-49 years in HIV care clinics for women in Kenya.

Specific Objectives I. Identify and address barriers to integration and uptake of cervical cancer screening and treatment linkage in HIV care settings in Kenya.

II. Evaluate the implementation and effectiveness of ENHANCE LINKage (HPV self-testing, care navigators, and mHealth that supports screening and treatment linkage) in a hybrid type 2 study, a cluster randomized trial in 20 HIV care clinics.

III. Evaluate sustainability and economic impacts of ENHANCE LINKage.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1 (PATIENTS): Aged 25-49 years
* AIM 1 (PATIENTS): Female
* AIM 1 (PATIENTS): Willing to participate in a 90-minute audio-recorded focus group discussion (FGD) and
* AIM 1 (PATIENTS): Speak English or Swahili
* AIM 1 (NURSES, CLINICAL STAFF, ADMINISTRATORS): Aged 18 years or older
* AIM 1 (NURSES, CLINICAL STAFF, ADMINISTRATORS): Involved in implementing intervention components
* AIM 1 (STAKEHOLDERS): Adults (aged >= 18 years) who are healthcare system users, support persons, healthcare providers and administrators, representatives of the government, professional associations, and non-governmental and faith-based organizations
* AIMS 2 AND 3 (CLINIC PROVIDERS): Aged 18 years and older involved in CC screening, triage, and treatment
* AIMS 2 AND 3 (WOMEN LIVING WITH HIV): Ages 25-49 years

Exclusion Criteria:

* AIM 1: Stakeholder Advisory Board (SAB) members who are not engaged in CC work, individuals who have recently retired from the selected clinics, and patients who are attending the clinic for the first time will be excluded from the study
* AIMS 2 AND 3 (WOMEN LIVING WITH HIV): Pregnant women, women =< 6 weeks postpartum, and women already confirmed to have cervical cancer will be excluded

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2280 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
IMPLEMENTATION OUTCOME: Difference in proportions in cervical cancer (CC) screening uptake between the intervention implementation versus control clinics | 1 to 12 months
  Modified mixed effects Poisson models will be used to estimate prevalence ratios, including the effect of clinic-level intervention (no intervention versus intervention) with fixed effects for intervention exposure status, and a random effect for clinic. Imbalanced baseline demographic and clinical characteristics across clinics will be included as independent variables in an adjusted model. Statistical differences between intervention versus control clinics during each observation period in terms of indicators will be tested using X^2 tests while mean differences and 95% confidence intervals (CI) will be tested using t-tests.
EFFECTIVENESS OUTCOME: Difference in the proportion of patients that received follow-up triage (with VIA) or treatment in the implementation intervention versus control clinics | 1 to 12 months
  Modified mixed effects Poisson models will be used to estimate prevalence ratios, including the effect of clinic-level intervention (no intervention versus intervention) with fixed effects for intervention exposure status, and a random effect for clinic. Imbalanced baseline demographic and clinical characteristics across clinics will be included as independent variables in an adjusted model. Statistical differences between intervention versus control clinics during each observation period in terms of indicators will be tested using X^2 tests while mean differences and 95% CI will be tested using t-tests.

SECONDARY OUTCOMES:
Communication of human papillomavirus (HPV) test result to patients via mobile (m)Health messages | 1 to 12 months
  Based on confirmation of HPV test results being sent to the participant's phone via two-way text message or mHealth application.
Receipt of HPV-negative result and guidance for next CC screening | 1 to 12 months
  Based on participants responding with a text to indicate that they have received their HPV results.
Retention in HIV Care (>=2 visits per year) | 1 to 12 months
  Between-arm comparison
HIV viral suppression (undetectable) | 1 to 12 months
  between-arm comparison

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chung, MD, PhD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Kenya Medical Research Institute, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Undecided
Depends on regulations in Kenya regarding IPD